CLINICAL TRIAL: NCT03907943
Title: Assessment of Cognitive Function in Patients Undergoing Elective Carotid Endarterectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Semmelweis University Heart and Vascular Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 17/2019
Record Dates: First submitted 2019-03-26; First posted 2019-04-09 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Endarterectomy, Carotid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical treatment of carotid endarterectomy (Other): The change in the cognitive function will be assessed in all patient undergoing carotid endarterectomy.
  Interventions: Procedure: carotid endarterectomy

INTERVENTIONS:
Procedure: carotid endarterectomy — Surgical treatment of ICA stenosis.

SUMMARY:
Assessment of cognitive function in patients undergoing elective carotid endarterectomy

Classical treatment for ICA stenosis is carotid endarterectomy (CEA), which has been proven effective in preventing future stroke as well as improving cerebral perfusion. However, the influence of CEA on cognition is less defined, it remains unclear whether CEA can improve cognitive function. A change in cognition is one of the most threatening diseases of recent years, cognitive impairment significantly impacts patients, families, and healthcare system.

The difference in the cognitive outcome may be accounted for microembolic events and adverse changes in haemodynamic circumstances.

The aim of our study is to identify those factors what may have role in the postoperative cognitive decline.

The study was approved by the Ethical Committee of the university ( SE RKEB: 17/2019) and written informed consent will be obtained from all patients.

The investigators intend to enroll patient aged more than 18 years undergoing elective carotid endarterectomy at our hospital ( Semmelweis University Heart and Vascular Center). Exclusion criterion included young age (less than 18 years), incapacity and urgent surgery. The investigators would like to register at least 100-150 patients in our study.

Most relevant anamnestic dates, the results of the laboratory and radiological reports will be recorded. Cognitive functions will be assessed one day before, one day and six month after the surgery using MMSE and a questionnaire called Frailty to characterize beside cognitive function the physiological reserve of the patients too.

The investigators manage patients undergoing carotid endarterectomy with general anaesthesia, using inhaled or total intravenous agents.

During the operation the investigators record beside the routine monitoring (intraarterial blood pressure, ECG, oxygen saturation, EtCO2, MAC) the cerebral tissue oxygen saturation using a near-infrared cerebral oximeter (Invos Cerebral/Somatic Oximeter) and the activity of the brain using GE Entropy Module.

The investigators would like to register the changes in the haemodynamic and cerebral condition and compare these results against the clinical outcome and the changes of the questionnaires.

Statistical analyses will be performed using Statistical Package for the Social Sciences.

ELIGIBILITY:
Inclusion Criteria:

* aged more than 18 years, undergoing elective carotid endarterectomy

Exclusion Criteria:

* younger than 18 years, incapacity, urgent surgery, lack of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients aged more than 18 years will be enrolled.
Enrollment: 150 (Estimated)
Dates: Start 2019-03-04 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive function after carotid endarterectomy | six months
  Change in MMSE score after the carotid endarterectomy compared to baseline.
Change in cognitive function after carotid endarterectomy | six months
  Change in Montreal Cognitive Assessment test after the endarterectomy compared to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Heart and Vascular Center, Budapest, Pest County, Hungary

IPD SHARING:
Plan to Share IPD: No